CLINICAL TRIAL: NCT00392496
Title: A Phase II Study of Sunitinib (SU11248; NSC 736511; IND 74019), an Oral Multi-Targeted Tyrosine Kinase Inhibitor, in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Sunitinib in Treating Patients With Relapsed or Refractory Diffuse or Mediastinal Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00692; NCI-2009-00692 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000652059; NCIC-182 (Other: National Cancer Institute of Canada Clinical Trials Group); NCIC-182 (Other: CTEP)
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Results first posted 2013-12-12 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2013-04

CONDITIONS: Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Sunitinib

ARMS (1):
- Arm I (Experimental): This is a non-randomized, open-label, multicenter study. Patients receive sunitinib malate orally once daily on days 1-28. Treatment repeats every 4 weeks for a maximum of 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate — Given orally
  Other Names: SU11248; sunitinib; Sutent

SUMMARY:
This phase II trial is studying how well sunitinib works in treating patients with relapsed or refractory diffuse or mediastinal large B-cell lymphoma. Sunitinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate in patients with relapsed or refractory, diffuse or mediastinal, large B-cell lymphoma treated with sunitinib malate.

II. Determine the toxicity of this drug in these patients. III. Determine the effects of this drug on peripheral blood biomarkers, circulating endothelial cells, and their precursors in these patients.

OUTLINE: This is a non-randomized, open-label, multicenter study.

Patients receive sunitinib malate orally once daily on days 1-28. Treatment repeats every 4 weeks for a maximum of 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
Criteria:

* Histologically confirmed diffuse or mediastinal large B-cell lymphoma*, meeting the following criteria: Advanced or metastatic disease, Incurable by standard therapies, Relapsed or refractory disease [Note: *Patients with diffuse large B-cell lymphoma whose disease has transformed from an earlier diagnosis of low grade lymphoma (i.e., an indolent histology) are eligible]
* Bidimensionally measurable disease** by CT scan, MRI, or physical exam, with >= 1 disease site meeting 1 of the following criteria: Lymph nodes >= 1.5 cm x 1.5 cm by spiral CT scan, Non-nodal regions >= 1 cm x 1 cm by MRI, CT scan, or physical exam [Note: **Bone lesions are not considered bidimensionally measurable disease]
* Received 1-2 prior chemotherapy regimens that included doxorubicin hydrochloride; Prior stem cell transplantation and high-dose chemotherapy is considered one regimen; One prior non-chemotherapy regimen in the form of radiation allowed; Measurable disease must be outside the previously irradiated area;
* No sole site of disease in a previously irradiated area unless progressive disease or new lesions are documented; Low-dose palliative radiotherapy may be allowed
* No known brain metastases
* Life expectancy >= 12 weeks
* ECOG performance status 0-1
* Absolute granulocyte count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* AST and ALT =< 2.5 times upper limit of normal (ULN)
* Bilirubin normal
* Calcium =< 3 mmol/L
* Creatinine =< 1.25 times ULN OR creatinine clearance >= 60 mL/min
* LVEF normal by MUGA
* None of the following in the past 12 months: cardiac arrhythmia, cerebrovascular accident (CVA), coronary/peripheral artery bypass graft or stenting, myocardial infarction, stable or unstable angina, symptomatic congestive heart failure, transient ischemic attack, pulmonary embolism
* No uncontrolled hypertension (systolic blood pressure >= 140 mm Hg or diastolic blood pressure >= 90 mm Hg)
* No New York Heart Association (NYHA) class III or IV heart disease
* No QTc prolongation (QTc interval >= 500 msec) or other significant ECG abnormalities
* No other prior malignancies except nonmelanoma skin cancer, in situ cervical cancer, or other solid tumors curatively treated with no evidence of disease for >= 5 years
* No history of allergic reaction to compounds of similar chemical or biological composition to sunitinib malate
* No other serious illness or medical condition that would preclude study participation, including, but not limited to, the following:

active, uncontrolled infection, serious or nonhealing wound, ulcer, or bone fracture, history of significant neurologic or psychiatric disorder that would impair the ability to obtain consent or limit compliance

* Other medical condition that might be aggravated by treatment
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No bowel obstruction
* No condition that would impair the ability to swallow and retain sunitinib malate tablets, including any of the following:

Gastrointestinal tract disease resulting in inability to take oral medication or a requirement for IV alimentation, Prior surgical procedures affecting absorption, Active peptic ulcer disease

* No pre-existing hypothyroidism unless euthyroid on medication
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* At least 28 days since prior chemotherapy
* At least 28 days since prior radiotherapy and recovered; radiotherapy must have involved < 30% of functioning bone marrow
* At least 28 days since prior major surgery and recovered
* At least 12 days since prior and no concurrent CYP3A4 inducers, including any of the following: rifampin, phenytoin, rifabutin, hypericum perforatum (St. John's wort), carbamazepine, efavirenz, phenobarbital, tipranavir,
* At least 7 days since prior and concurrent CYP3A4 inhibitors, including any of the following: azole antifungals (e.g., ketoconazole, itraconazole), verapamil, clarithromycin, HIV protease inhibitors (e.g., indinavir, saquinavir, ritonavir, atazanavir, nelfinavir), erythromycin, delavirdine, diltiazem,
* No prior therapy with other antiangiogenic agents or multitargeted tyrosine kinase inhibitors, including any of the following:

bevacizumab, sorafenib tosylate, pazopanib, thalidomide, AZD2171 vandetanib, AMG 706, vatalanib, VEGF Trap

* No concurrent therapeutic doses of coumarin-derivative anticoagulants (e.g., warfarin); Concurrent dosing of =< 2 mg of warfarin daily for prophylaxis of thrombosis is allowed; Concurrent low molecular weight heparin is allowed provided INR is =< 1.5
* No other concurrent anticancer treatments, including investigational agents
* No concurrent agents with proarrhythmic potential, including any of the following: terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide, flecainide
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rena Buckstein, Principal Investigator — Canadian Cancer Trials Group
Locations (1):
- National Cancer Institute of Canada Clinical Trials Group, Kingston, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was centrally activated on November 8, 2006 and closed to accrual on March 24, 2009. Patients were recruited from 5 cancer centres in Canada
Period: Overall Study
Arm/Group | Arm I
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Two patients who were determined as ineligible were excluded from all analyses
Arm/Group | Arm I
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 65 [34 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Region of Enrollment [Number; unit: participants]
  Canada | 17

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response
Description: It is defined as per the Report of the International workshop to standardize response criteria for non-Hodgkin's lymphoma and reviewed independently
Time Frame: Up to 3 years
Population: patients evaluable for response
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 15
participants | 0

ADVERSE EVENTS:
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 13/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=17)
Grade 2 somnolence (Nervous system disorders) | 1
Grade 2 Hypothyroidism (Investigations) | 1
Grade 2 Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1
Grade 4 fatigue (General disorders) | 1
Grade 3 ALT, gr 2 AST and gr 2 alkaline phosphatase (Investigations) | 1
Hospitalization for gr 4 platelets and gr 3 hemoglobin (Investigations) | 1
Grade 3 AST (Investigations) | 1
Death not associated with CTCAE term (General disorders) | 3
Grade 2 dysphagia and hypothyroidism (Gastrointestinal disorders) | 1
Grade 2 Rigors/chills (General disorders) | 1
Hospitalization for Grade 3 dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hospitalization for grade 3 GI Bleed (Gastrointestinal disorders) | 1
Hospitalization for infected lymphoma lesion (skin: cellulitis grade 5) (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=17)
Supraventricular arrhythmia Sinus tachycardia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 4
Hypotension (Cardiac disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Fatigue (General disorders) | 14
Fever (General disorders) | 4
Insomnia (General disorders) | 3
Rigors/chills (General disorders) | 2
Sweating (General disorders) | 2
Decubitus (Skin and subcutaneous tissue disorders) | 1
Hand-foot (Skin and subcutaneous tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Anorexia (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 9
Dehydration (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 8
Distension (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Heartburn (Gastrointestinal disorders) | 8
Mucositis (clinical exam) Oral cavity (Gastrointestinal disorders) | 4
Mucositis (functional/symptomatic) Oral cavity (Gastrointestinal disorders) | 4
Mucositis (functional/symptomatic) Pharynx (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Taste alteration (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 7
GI - Other (Gastrointestinal disorders) | 2
Hemorrhage pulmonary Nose (Blood and lymphatic system disorders) | 3
Hemorrhage, GI Oral cavity (Blood and lymphatic system disorders) | 1
Hemorrhage, GI Stomach (Blood and lymphatic system disorders) | 1
Infection with normal ANC Bladder (Infections and infestations) | 1
Infection with normal ANC Lung (Infections and infestations) | 1
Infection with normal ANC Pelvis NOS (Infections and infestations) | 1
Infection with normal ANC Skin (Infections and infestations) | 1
Infection with normal ANC Upper airway NOS (Infections and infestations) | 1
Infection with unknown ANC Blood (Infections and infestations) | 1
Infection with unknown ANC Lip/perioral (Infections and infestations) | 1
Infection - Other (Infections and infestations) | 1
Edema: limb (Blood and lymphatic system disorders) | 4
Lymphatics - Other (Blood and lymphatic system disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Gait/walking (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1
Confusion (Nervous system disorders) | 1
Mood alteration Anxiety (Nervous system disorders) | 1
Mood alteration Depression (Nervous system disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 7
Somnolence (Nervous system disorders) | 1
Diplopia (Eye disorders) | 1
Pain Abdomen NOS (General disorders) | 6
Pain Back (General disorders) | 5
Pain Bladder (General disorders) | 1
Pain Bone (General disorders) | 1
Pain Chest/thorax NOS (General disorders) | 1
Pain Extremity-limb (General disorders) | 3
Pain Head/headache (General disorders) | 3
Pain Joint (General disorders) | 3
Pain Lymph node (General disorders) | 1
Pain Middle ear (General disorders) | 1
Pain Muscle (General disorders) | 2
Pain Oral cavity (General disorders) | 4
Pain Pain NOS (General disorders) | 1
Pain Tumor pain (General disorders) | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (General disorders) | 6
Dyspnea (General disorders) | 8
Pleural effusion (General disorders) | 2
Voice changes (General disorders) | 2
Pulmonary - Other (General disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less